CLINICAL TRIAL: NCT03431506
Title: Vestibular Function and Vestibular Rehabilitation in Sudden Sensorneural Hearing Loss With Vertigo
Brief Title: Vestibular Function and Vestibular Rehabilitation in SSHL With Vertigo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Vestibular function in SSHL
Record Dates: First submitted 2018-01-16; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Vestibular Disorder
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-training group (Active Comparator)
  Interventions: Behavioral: Vestibular rehabilitation
- training group (Experimental)
  Interventions: Behavioral: Vestibular rehabilitation

INTERVENTIONS:
Behavioral: Vestibular rehabilitation — Vestibular Rehabilitation Exercises

SUMMARY:
To evaluate the vestibular function and vestibular rehabilitation in sudden sensorneural hearing loss(SSHL) with vertigo

DETAILED DESCRIPTION:
Approximately 5-20 per 100,000 persons are afflicted with SSHL annually, and nearly 20-60% of SSHL patients complain of simultaneous vertigo.The aim of this study was to evaluate the prevalence of vestibulocochlear lesions in sudden sensorneural hearing loss(SSHL) with vertigo, as well as the role of vestibular rehabilitation in the prognosis of SSHL with vertigo.

ELIGIBILITY:
Inclusion Criteria:

1. A rapid onset sensorineural hearing loss of more than 30 dB for at least three contiguous audiometric frequencies within a period of 3 days, according to standard AAO - HNS;
2. Within 10 days from onset;
3. Without other virus infectious disease within three months.

Exclusion Criteria:

1. BPPV; Meniere's disease and vestibular migraine.
2. With certain Known etiology, including acoustic neuroma, heart cerebrovascular accident, injury, Hunt syndrome, etc

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of vestibular function status by vestibular function tests in SSHL with vertigo at stage 1(before treatment) | before treatment
  Vestibular function status in SSHL with vertigo at stage 1(before treatment)

SECONDARY OUTCOMES:
Assessment of vestibular function status by vestibular function tests in SSHL with vertigo at stage 2(2 weeks after treatment) | 2 weeks after treatment
  Vestibular function status in SSHL with vertigo at stage 2(2 weeks after treatment)
Assessment of vestibular function status by vestibular function tests in SSHL with vertigo at stage 2(2 months after treatment) | 2 months after treatment
  Vestibular function status in SSHL with vertigo at stage 2(2 months after treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Otorhinolaryngology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No